CLINICAL TRIAL: NCT05728190
Title: Effect of Inhalation Aromatherapy on Pain, Anxiety, and Sleep Quality in Burn Patients
Brief Title: Effect of Aromatherapy on Pain, Anxiety and Sleep Quality in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sema Koçaşlı (Other)
Responsible Party: Sponsor-Investigator, Sema Koçaşlı, Assist. Prof. Dr., Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1929/2021
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Aromatherapy
Keywords: burn; Anxiety; lavender aromatherapy; nursing; pain; sleep quality
MeSH Terms: conditions — Burns; Anxiety Disorders; Pain; Sleep Initiation and Maintenance Disorders | interventions — lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender essential oil (Experimental): In the intervention group, five days, seven drops of lavender essential oil were dripped onto a 5x5 gauze pad in the morning and evening, for 20 minutes, 10 cm away from the nose, and sniffed.
  Interventions: Other: Lavender essential oil
- Steril/Salin water (Placebo Comparator): Five days seven drops of saline/sterile water were dripped onto a 5x5 gauze pad in the morning and evening, and they were put to sniff for 20 minutes, 10 cm away from the nose.
  Interventions: Other: steril/salin water

INTERVENTIONS:
Other: steril/salin water — Five days seven drops of saline/sterile water were dripped onto a 5x5 gauze pad in the morning and evening, and they were put to sniff for 20 minutes, 10 cm away from the nose. Green food coloring was added (one drop of food coloring to 5 ml of sterile/saline water) to make sterile/saline water similar to lavender oil.
  Arms: Steril/Salin water
Other: Lavender essential oil — Five days seven drops of lavender essential oil were dripped onto a 5x5 gauze pad in the morning and evening, for 20 minutes, 10 cm away from the nose, and sniffed.
  Arms: Lavender essential oil

SUMMARY:
This study, which was designed as a randomized placebo-controlled experimental study, was conducted to determine the effect of inhalation aromatherapy with lavender essential oil on pain, anxiety and sleep quality in burn patients.

DETAILED DESCRIPTION:
After 5 patients were included in the sample size of the study, intervention and control groups, power analysis was performed using the G*Power Software (3.1.9.2) program. With a margin of error of 5%, an effect size of 0.15, and a power of 95%, the sample group size was calculated as 54 patients. Considering that data loss might be 10% on average in the study, it was decided to recruit 60 patients. Participants were randomized according to patient rooms. There are a total of 11 rooms and 16 beds in the burn unit, 5 double and 6 single. 11 rooms are numbered sequentially according to their location in the corridor.

In the intervention group, seven drops of lavender essential oil were dripped onto a 5x5 gauze pad in the morning and evening, for 20 minutes, 10 cm away from the nose, and sniffed.

In the placebo control group, seven drops of saline/sterile water were dripped onto a 5x5 gauze pad in the morning and evening, and they were put to sniff for 20 minutes, 10 cm away from the nose. Green food coloring was added (one drop of food coloring to 5 ml of sterile/saline water) to make sterile/saline water similar to lavender oil. Data were collected using Individual Data Collection Form, Spielberg State Anxiety Scale, Visual Analog Scale, Richard Campbell Sleep Scale before and after five days of morning and evening aromatherapy application.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* 2nd and/or 3rd degree burns but not in emergency/resuscitative phase,
* Total body burn area is 5-30%,
* No acute-chronic respiratory system disease (asthma, COPD, etc.),
* No problem in sense of smell,
* No communication problem,
* Not participating in another study at the same time,
* Patients who volunteered to participate in the study.

Exclusion Criteria:

* Those who are allergic to lavender essential oil,
* Having a history of head trauma or convulsions,
* Having respiratory tract (inhalation) burn,
* Having alcohol or narcotic substance addiction,
* Having a history of pregnancy, epilepsy, high blood pressure and migraine,
* Patients undergoing intubation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 5 days
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Spielberg State Anxiety Scale | 5 days
  The scale has a four-point Likert structure consisting of 20 items and a total score of 20-80 is obtained.
  A score of 20 or less indicates that the individual does not have anxiety, a score between 21-39 indicates mild anxiety, a score between 40-59 indicates moderate, and a score between 60-80 indicates a high level of anxiety.
Richard Campbell Sleep Scale | 5 days
  There are 6 items in the scale. There are 5 items in the assessment. Each item is evaluated on the scale between 0 and 100. If the score is between "0-25", it indicates very bad sleep, and between "76-100" indicates very good sleep.

CONTACTS AND LOCATIONS:
Overall Officials: ayten akkaya, PhD, Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Ankara Medipol University, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No